CLINICAL TRIAL: NCT00186784
Title: Repetitive Transcranial Magnetic Stimulation (rTMS) in Unipolar Depression
Brief Title: Transcranial Magnetic Treatment (TMS) in Unipolar Depression
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: Queen's University, Kingston, Ontario (Other)
Responsible Party: Dr. Gary M. Hasey, St. Joseph's Healthcare
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: TMS1871
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2011-08-03 (Estimated); Status verified 2011-08

CONDITIONS: Unipolar Depression
Keywords: Repetitive Transcranial Magnetic Stimulation; TMS
MeSH Terms: conditions — Depressive Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Transcranial Magnetic Stimulation (TMS) — treatment for 10 days

SUMMARY:
Repetitive Transcranial Magnetic Stimulation (rTMS) can improve mood and decrease sadness in patients with depression.

In this study, the investigators seek to increase their understanding about how rTMS improves depression, and to determine which form of rTMS is most effective for depression, when used in combination with antidepressant medication.

DETAILED DESCRIPTION:
Patients will be assigned for 4 treatment arms, receiving either left high frequency plus right low frequency, or left high frequency plus right sham, or left sham, plus right low frequency, or left sham plus right sham treatment. All subjects will receive treatments for 10 days and will be followed for another 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Major Depression
* No physical health problems

Exclusion Criteria:

* History of Epilepsy
* Metal in the head/neck or skull
* Pacemaker
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2000-12; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale | Pre TMS and post TMS
Beck Depression Rating Scale | pre TMS and post TMS

SECONDARY OUTCOMES:
Quantitive Electroencephalographic(QEEG)activity and measures of regional cerebral blood flow | pre TMS and post TMS as well as post phase II, second set of TMS

CONTACTS AND LOCATIONS:
Overall Officials: Gary Hasey, MD, Principal Investigator — McMaster University
Locations (1):
- St.Joseph's Healthcare, rTMS Laboratory, Mood Disorders Program, 100 West Fifth Street, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Jacquot F, Khoury S, Labrum B, Delanoe K, Pidoux L, Barbier J, Delay L, Bayle A, Aissouni Y, Barriere DA, Kultima K, Freyhult E, Hugo A, Kosek E, Ahmed AS, Jurczak A, Lingueglia E, Svensson CI, Breuil V, Ferreira T, Marchand F, Deval E. Lysophosphatidylcholine 16:0 mediates chronic joint pain associated to rheumatic diseases through acid-sensing ion channel 3. Pain. 2022 Oct 1;163(10):1999-2013. doi: 10.1097/j.pain.0000000000002596. Epub 2022 Jan 27. PMID 35086123